CLINICAL TRIAL: NCT05916651
Title: The PRYME Study: Promoting Resilience in Youth Through Mindfulness mEditation.
Brief Title: Promoting Resilience in Youth Through Mindfulness mEditation
Acronym: PRYME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Donders Centre for Cognitive Neuroimaging (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL82568.091.22; 60-63600-98-1054 (Other Grant/Funding Number: Netherlands Organisation for Health Research and Development); 29875 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2023-05-30; First posted 2023-06-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-07

CONDITIONS: Internalizing Problems
Keywords: mindfulness; internalizing problems; self-referential processing; youth; help-seeking; resilience

STUDY DESIGN:
Intervention Model Description: The PRYME study is a Randomized Controlled Trial (RCT) that compares care-as-usual (e.g., supportive counseling by a student psychologist or mental health nurse-practitioner) with care -as-usual + mindfulness training. Participants are randomized to either of these conditions. Data is collected at baseline, after the mindfulness training (approximately 3 months after baseline), and at 2 and 6 months follow-up. Multiple measurements will be conducted using questionnaires, experimental tasks in and out of the MRI scanner, MRI scans, and clinical interviews.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (LOS training) + care as usual (intervention group) (Experimental): Intervention group: mindfulness (LOS) training + CAU
  Interventions: Behavioral: Learning to Offset Stress (LOS) (in Dutch: Leren Omgaan met Stress) training; Behavioral: Care as usual
- Care-as-usual (CAU)-only (control group) (Active Comparator): Control group: CAU-only
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Learning to Offset Stress (LOS) (in Dutch: Leren Omgaan met Stress) training — The investigational treatment is the LOS training, which is an adaptation of two previously validated mindfulness-based programs: Mindfulness-Based Cognitive Therapy (MBCT) developed by Segal, Williams, and Teasdale (2002) and the Mindful2Work (M2W) program developed by de Bruin, Formsma, and Bögels (2018). The M2W program combines mindful physical activity, yoga, and mindfulness meditation to target stress symptoms and burn-out in adults. The LOS training was adapted from these programs to meet the needs of youth with internalizing problems. The training consists of 8 weekly 2-hour sessions that each comprise three elements: mindful physical activity (15-20 minutes), yoga (15-20 minutes), and mindfulness meditation exercises (80-90 minutes). In addition to attending group sessions, participants are invited to practice at home on a daily basis. Home practice consists of daily mindfulness practices comprising mindfulness exercises, yoga and mindful physical activity.
  Arms: Intervention (LOS training) + care as usual (intervention group)
Behavioral: Care as usual — Youth who seek help for internalizing problems from a primary mental health practitioner, including student psychologists or mental health nurse practioners, but do not (yet) meet criteria for (major) mental illness are typically offered supportive counselling, aimed primarily at helping people feel understood and supported. Supportive counselling may also include instructions on behavioral activation, particularly when individuals report reduced activity and behavioral avoidance including social withdrawal. In addition, mental health practitioners commonly employ a "watchful waiting" policy for people with symptoms in the milder range, where they check-in with clients on a regular basis and refer for more intensive treatment if and when symptoms worsen.

SUMMARY:
The aim of this randomized controlled trial (RCT) is to assess whether mindfulness training reduces early stage internalizing problems such as anxiety, worrying, and low mood in help-seeking youth.

Participants will be randomly assigned to one of two groups: 1) mindfulness + care-as-usual (CAU) or 2) CAU-only. The mindfulness program was developed specifically for youth with internalizing problems. The 8-week training program consists of weekly 2-hour sessions, with mindfulness, yoga, and mindful active movement in each session. In addition, participants are invited to practice at home in between sessions for around 20 minutes per day.

Data will be collected at baseline (T0), end-of-treatment (T1) (or 2-3 months after baseline for the CAU-only group), and at 2 months follow-up (T2) and 6 months follow-up (T3).

Measurements will include:

* Self-report questionnaires (T0, T1, T2, T3)
* Psychiatric diagnostic interview (T0, T3)
* MRI scans (T0, T1)
* Cognitive tasks (T0, T1)

The primary outcome parameter is the total number of internalizing problems measured with the Adult Self Report (ASR) at end-of-treatment. The effect of mindfulness training (mindfulness + CAU vs. CAU-only) on internalizing problems at T1 will be assessed using a linear-mixed effects model.

DETAILED DESCRIPTION:
The main aim of this study is to assess whether mindfulness training reduces early-stage mental problems such as anxiety, worrying, and low mood in help-seeking youth.

Background The majority of mental illnesses (75%) emerge before the age of 25 and many have a life-long impact on health and functioning. Early intervention may be more effective than treatment required in later stages. The early stage of mental illness is typically characterized by mild, non-specific complaints such as anxiety, worrying, and low mood. These "internalizing problems" are increasingly common in youth and associated with various adverse outcomes including mental illness development and therefore represent an important target for early intervention.

Internalizing problems are observed in the early stages of various mental disorders. Help-seeking youth with internalizing problems may thus reflect an early stage of mental illness development. Mindfulness training is effective in the treatment of a range of mental disorders including major depression and may promote resilience by acting on underlying mechanisms. In mindfulness training, participants learn to focus and sustain attention on present-moment experiences in a non-judgmental manner. This process fosters awareness of automatic patterns of behavior and improves cognitive flexibility and emotion regulation.

Research shows that a network of brain regions involved in the processing of self-related information (i.e., Default Mode Network; DMN) is hyperactive in people with serious mental illness. Individuals who are at risk for depression are prone to interpret experiences in a negative, self-critical manner. MRI studies have shown that mindfulness reduces activity of the DMN during processing of self-relevant information. Mindfulness training may thus normalize abnormalities in self-referential processing and thereby reduce risk of mental illness development.

Study design This study is a Randomized Controlled Trial. Participants are randomly assigned to one of two groups: 1) the intervention group, who receives mindfulness training in addition to care-as-usual (CAU) and 2) the control group, who receives CAU-only. Research team members who perform clinical follow-up assessments are blind to group-allocation. Data is collected at 4 time points: baseline (T0), end-of-treatment (T1) (within 1 month after completing the mindfulness training intervention group, and approximately 3 months after the baseline measurement for the control group), 2-months follow-up (T2), and 6-months follow-up (T3). Assessments include clinical interviews, self-report questionnaires, and cognitive tasks and MRI scans (at baseline and end-of-treatment only). The main outcome is the total number of internalizing problems at T1 as measured with the Adult Self Report (ASR). Secondary data include self-report questionnaires on comorbid symptoms, rumination, self-esteem, experiential avoidance, mindfulness skills, self-compassion, social and emotional well-being and resilience.

MRI and experimental task data are acquired to assess (changes in) underlying neurocognitive mechanisms and neural correlates. MRI scans are acquired at baseline and T1 and include an anatomical scan, diffusion-MRI scan, and resting-state fMRI scan. In addition, the Self-Referent Encoding Task (SRET), which measures biases for positive and negative self-related information, is acquired in the scanner. Furthermore, participants perform an aversive go/no-go task to measure escape/avoidance behavior in the context of aversive cues. In addition, participants are invited to perform a Pavlovian-to-Instrumental Transfer (PIT) task and Control Belief Updating (CBU) task online. The PIT task measures how Pavlovian biases influence instrumental approach and withdrawal behavior. The CBU measures the extent to which one can flexibly update beliefs about the controllability of their environment.

Study population Help-seeking youth (16-25 years of age) will be recruited from primary (mental) health care providers, including student psychologists, general practitioners (GPs), and mental health nurse practitioners. As both internalizing problems and interest in mindfulness training are more common in women, an imbalance in sex (more women than men) is accepted. Sample size calculations to ensure adequate power to detect small to medium-sized group-differences in internalizing problems from baseline to T1, resulted in a required sample size of N = 155.

Interventional treatment The mindfulness program used in the study is the Learning to Offset Stress (LOS; in Dutch: Leren Omgaan met Stress) program. This 8-week mindfulness training program was designed specifically for youth with internalizing problems. The program consists of weekly 2-hour sessions, with mindfulness exercises, yoga and mindful physical activity in each session, and daily at-home practice (~20 min).

Care-as-usual Care-as-usual comprises all care from primary mental health care providers or secondary mental health services following referral. Primary mental health care typically involves supportive counseling and/or behavioral activation.

Nature and extent of the burden and risks associated with participation The risks and discomfort associated with participation in this study are estimated as low. The main burden consists of repeated non-invasive assessments and MRI scanning, which may be uncomfortable for some participants.

Hypothesis The main hypothesis is that mindfulness training + CAU relative to CAU-only will reduce internalizing problems at T1 as measured with the ASR.

Hypotheses on cognitive and MRI data will be described in detail elsewhere (aspredicted.com). Briefly, it is hypothesized that higher internalizing problems at baseline will be associated with higher negativity bias in endorsement and recall of self-related information on the SRET, exaggerated escape and avoidance responses on the aversive go/no-go task, increased aversive Pavlovian influence over instrumental behavior on the PIT, and a bias towards reduced controllability on the CBU task and that these effects will be attenuated following mindfulness training (+CAU) as compared to CAU-only.

ELIGIBILITY:
Inclusion Criteria:

1. Youth between 16 and 25 years of age
2. Provide written informed consent
3. Adequate mastery of Dutch language

Exclusion Criteria:

1. Lifetime diagnosis of severe major depression, bipolar disorder, schizophrenia spectrum disorder, personality disorder, and post-traumatic stress disorder
2. History of major medical illness or neurological illness
3. Participation in a mindfulness programme in the past year
4. Current participation in another intervention study
5. Moderate to severe substance use disorders (i.e., we will allow for mild substance use)
6. Current active suicidality, current psychotic symptoms above clinical cut-off for psychosis, or current trauma-related complaints above clinical cut-off for PTSD.
7. Diagnosed or suspected (mild) intellectual disability (estimated IQ < 75)

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The total number of internalizing problems as measured with the ASR, computed as the sum of responses on the items comprising withdrawn, somatic complaints, anxiety and depression subscales. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The ASR is a 126-item self-report questionnaire assessing aspects of adaptive functioning and problems. Items are rated on a 3-point scale: 0-Not True, 1-Somewhat or Sometimes True, 2-Very True or Often True.

SECONDARY OUTCOMES:
Presence of psychiatric disorders as per DSM-5 criteria on the MINI - Simplified for DSM-5 (MINI-S-DSM-5). Of note: the MINI-S is a separate instrument from the Mini Neuropsychiatric Interview (MINI) for DSM-5 by Prof. Sheehan. | 6-months follow-up (T3), approximately 9 months after the baseline assessment
  The MINI-S-DSM-5 is a structured diagnostic interview for psychiatric disorders, which assesses 16 common psychiatric disorders.
The Ruminative-Reflection Questionnaire (RRQ) - brooding subscale score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The RRQ is used to measure two factors of self-focused attention: rumination and reflection). The brooding subscale consists of 12 items that are measured on a 5-point Likert scale.
The Perceived Stress Scale (PSS-10) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The Perceived Stress Scale (PSS-10) is a self-report questionnaire measuring (perceived) stress. It consists of 10 items that are measured using a 4-point Likert scale. Total score ranges from 0-40.
The Rosenberg Self-Esteem Scale (RSES) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The RSES is a self-report questionnaire that assesses global self-esteem. It consists of 10 items that are measured using a 4-point Likert scale.
The Adaptive Self-Concept Questionnaire (ASCQ) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The ASCQ is a self-report questionnaire that measures properties of the self-concept that are associated with adaptability. It consists of 25 items that are measured using a 6-point Likert scale.
The Acceptance and Action Questionnaire (AAQ) total score | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The AAQ is a self-report questionnaire that measures experiential avoidance. It consists of 10 items that are measured using a 7-point Likert scale.
The Five Facets of Mindfulness Questionnaire - Short Form (FFMQ - SF) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The Five Facets of Mindfulness Questionnaire - Short Form (FFMQ - SF) is a self-report questionnaire that measures mindfulness skills. It consists of 24 items that are measured using a 5-point Likert scale.
The Self-Compassion Scale (SCS) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The Self-Compassion Scale (SCS) is a self-report questionnaire that measures self-compassion. It consists of 24 items that are measured using a 7-point Likert scale.
The Mental Health Continuum - Short Form (MHC - SF) total score | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The MHC - SF is a self-report questionnaire that measures social and emotional well-being. It consists of 14 items that are measured using a 6-point Likert scale.
The Connor-Davidson Resilience Scale (CD - RISC) total score. | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The CD - RISC is a self-report questionnaire that measures resilience. It consists of 10 items that are measured using a 5-point Likert scale.
Self-Referent Encoding Task (SRET) | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The SRET is a behavioral task that measures implicit biases for positive and negative self-related information. It will be partly conducted in the MRI scanner.
Escape/avoidance learning task | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The escape/avoidance learning task is an aversive go/no-go task. This task measures automated escape and avoidance behaviors in the context of aversive cues.
Pavlovian to Instrumental Transfer (PIT) task | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The PIT-task is a behavioral task that measures the influence of positive and negative Pavlovian biases on instrumental approach of withdrawal behavior. This task is performed online and is an optional part of the assessments for the participant.
Control Belief Updating (CBU) task | end-of-treatment (T1), approximately 3 months after the baseline assessment
  The CBU task is a behavioral task that measures the ability to flexibly update beliefs about environmental controllability. This task is performed online and is an optional part of the assessments for the participant.
MRI scanning | end-of-treatment (T1), approximately 3 months after the baseline assessment
  MRI scanning will include an anatomical scan (MPRAGE), resting state fMRI scan, diffusion-weighted MRI scan, and task-fMRI (SRET)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboud university medical center (Radboudumc), Nijmegen, Gelderland
  - Donders Centre for Cognitive Neuroimaging (DCCN), Nijmegen, Gelderland

REFERENCES:
- [Derived] Schepers M, Lagerweij P, Geurts D, Krause F, Ouden HD, Cools R, Speckens A, Collin G. Promoting Resilience in Youth through Mindfulness mEditation (PRYME): Study protocol for a randomized controlled trial investigating the effects of mindfulness training as add-on to care-as-usual on internalizing problems, mental illness development, and associated brain and cognitive processes in help-seeking youth. BMC Psychiatry. 2025 Feb 14;25(1):126. doi: 10.1186/s12888-024-06430-7. PMID 39948492